CLINICAL TRIAL: NCT00950859
Title: A Pilot Study to Assess the Antiviral Activity of GSK1349572 Containing Regimen in Antiretroviral Therapy (ART)-Experienced, HIV-1-infected Adult Subjects With Raltegravir Resistance
Brief Title: A Pilot Study Assessing the Integrase Inhibitor GSK1349572 in HIV-infected Persons With Virus Resistant to Raltegravir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112961
Record Dates: First submitted 2009-07-23; First posted 2009-08-03 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-09

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: treatment experienced; HIV Infection; raltegravir resistance; GSK1349572; optimized background regimen; integrase inhibitor
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1349572 Cohort I (Experimental): Single Arm, Cohort I
  Interventions: Drug: GSK1349572 (Cohort I)
- GSK1349572 Cohort II (Experimental): Single Arm, Cohort II
  Interventions: Drug: GSK1349572 (Cohort II)

INTERVENTIONS:
Drug: GSK1349572 (Cohort I) — 50 mg once daily
  Other Names: Dolutegravir
  Arms: GSK1349572 Cohort I
Drug: GSK1349572 (Cohort II) — 50 mg twice daily
  Other Names: Dolutegravir
  Arms: GSK1349572 Cohort II

SUMMARY:
Integrase is an enzyme produced by HIV so that the virus can multiply in the human body. GSK1349572 is a new drug in the integrase inhibitor class that prevents the enzyme from working properly and therefore prevents the virus from multiplying.

GSK1349572 has shown to be effective against viruses in a short-term monotherapy study in adults with no previous exposure to integrase inhibitors. The purpose of this study is to determine whether GSK1349572 is effective in the treatment of HIV-infected patients who no longer respond to treatment with the approved integrase inhibitor raltegravir and carry viruses with resistance to this drug. The safety and efficacy of GSK1349572 50mg once daily in combination with the background HIV drugs previously administered (unless discontinuation of a particular drug is required) will be assessed over 10 days (functional monotherapy phase), followed by the evaluation of the safety and efficacy of GSK1349572 given with a new optimised background regimen from Day 11 through at least Week 24.

DETAILED DESCRIPTION:
Study (ING112961) is a Phase IIb, multicentre, open-label, single arm, two cohorts, pilot study to assess the antiviral activity of GSK1349572 containing regimen in HIV-1 infected ART-experienced adults with raltegravir (RAL) resistance. The study will include approximately 50 ART-experienced subjects with either current or past virologic failure to RAL. All subjects must harbour isolates with RAL resistance mutations at Screening. Subjects should also have documented genotypic and/or phenotypic resistance to at least one compound from each of three or more of the approved classes of ART (including integrase inhibitors [INIs]). Subjects with current RAL virologic failure will substitute RAL with GSK1349572 50mg once daily and continue the remaining components of their failing regimen through Day 10. Subjects with historical RAL virologic failure will add GSK1349572 50mg once daily to their failing regimen through Day 10. On Day 11 all subjects will continue GSK1349572 and optimize their background therapy. Antiviral activity, safety and tolerability of GSK1349572 will be evaluated at Day 11 and over time through at least Week 24.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected male or female adults at least 18 years of age with a plasma HIV-1 RNA > 1,000 copies/mL at study entry. Women capable of becoming pregnant must use appropriate contraception during the study (as defined by the protocol)
* ART-experienced (defined as on stable ART for at least the last 2 months) and is either currently experiencing virologic failure to RAL or experienced virologic failure to RAL > 8 weeks prior to Screening
* Must have documented RAL genotypic resistance on study entry genotype
* Must have documented genotypic or phenotypic resistance to at least one drug from each of three or more of all approved classes of ART
* For Cohort II, Subjects MUST be able to receive at least one fully active drug as part of the Day 11 optimised background regimen
* Willing and able to understand and provide signed and dated written informed consent prior to screening

Exclusion Criteria:

* Any pre-existing mental, physical, or substance abuse disorder which, which could compromise ability to comply with the protocol or compromise subject safety
* Women who are pregnant or breastfeeding
* An active AIDS-defining condition at the screening visit
* Currently take and/or anticipated need for EFV, NVP, FPV/RTV or TPV/RTV during the study
* Treatment with any of the following medications within 15 days of starting study drug, or anticipated to need, during the course of the study: Etravirine (unless co-administered with LPV/RTV or DRV/RTV), rifampin, rifabutin, phenytoin, phenobarbital, barbiturates, glucocorticoids, modafinil, oxcarbazepine, pioglitazone, troglitazone, carbamazepine, St. Johns wort
* Previous participation in an experimental drug and/or vaccine trial(s) within 30 days or 5 half-lives
* History of ongoing or clinically relevant pancreatitis or hepatitis within the previous 6 months
* Expected to require treatment for HCV infection during the first 24 weeks of the study
* Evidence of cirrhosis with or without hepatitis viral co-infection
* History of upper gastrointestinal bleed and/or active peptic ulcer disease
* Screening haemoglobin <10g/dL (100g/L)
* Subject suffers from a serious medical condition which could compromise the safety of the subject.
* Any condition that could interfere with the absorption, distribution, metabolism or excretion of the drug or render the subject unable to take oral medication
* Screening lipase 3 times the upper limit of normal (ULN)
* Any acute or Grade 4 laboratory abnormality at screening
* Screening alanine aminotransferase (ALT) >5xULN
* Screening ALT 3xULN and bilirubin 1.5xULN (with 35% direct bilirubin)
* Personal or family history of prolonged QT syndrome.
* Any clinically significant finding, as specified in the protocol, on screening or baseline electrocardiograph (ECG)
* History of allergy to the study drugs or their components or drugs of their class
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days prior to screening, or future need of treatment with these agents during the study
* Treatment with immunomodulators within 28 days prior to screening or subject has received an HIV-1 vaccine within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (25):
- United States (11):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Dallas, Texas
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (7):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
- GSK Investigational Site, Milan, Lombardy, Italy
- Spain (4):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville

REFERENCES:
- [Background] Eron JJ, Clotet B, Durant J, Katlama C, Kumar P, Lazzarin A, Poizot-Martin I, Richmond G, Soriano V, Ait-Khaled M, Fujiwara T, Huang J, Min S, Vavro C, Yeo J; VIKING Study Group. Safety and efficacy of dolutegravir in treatment-experienced subjects with raltegravir-resistant HIV type 1 infection: 24-week results of the VIKING Study. J Infect Dis. 2013 Mar 1;207(5):740-8. doi: 10.1093/infdis/jis750. Epub 2012 Dec 7. PMID 23225901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited initially to Cohort I and subsequently to Cohort II. Recruitment to Cohort I was closed 9 months before recruitment to Cohort II was opened. Recruitment was not randomized.
Groups:
- Cohort I (DTG 50 mg OD): Participants received dolutegravir (DTG) 50 milligrams (mg) once a day (OD).
- Cohort II (DTG 50 mg BID): Participants received DTG 50 mg twice a day (BID).
Period: Overall Study
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Started | 27 | 24
Completed | 11 | 14
Not Completed | 16 | 10
Not completed — Adverse Event | 3 | 3
Not completed — Insufficient Viral Load Response | 12 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID) | Total
Number analyzed (Participants) | 27 | 24 | 51
Age, Customized [Median (Full Range); unit: Years]
  Years | 48 [19 to 61] | 47 [33 to 68] | 47 [19 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 25 | 18 | 43
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3 | 5 | 8
  White-Arabic/North African Heritage | 1 | 1 | 2
  White-White/Caucasian/European Heritage | 23 | 18 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved HIV-1 RNA <400 Copies (c)/Milliliter (mL) or at Least 0.7 log10 c/mL Below Their Baseline Value at Day 11
Description: The number of participants who acheived Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) <400 c/mL or at least 0.7 log10 c/mL below their Baseline value at Day 11 was assessed. The last observation was carried forward if a participant had missed the Day 11 visit. The Baseline observation was carried forward if a participant had discontinued the treatment before Day 11. Blood samples for assessment of HIV-1 RNA levels were collected at Baseline and Day 11.
Time Frame: Baseline (Day 1) and Day 11
Population: Intent-to-Treat Exposed (ITT-E) Population: all participants who received at least one dose of study medication and who had at least one post-Baseline measure of plasma HIV-1 RNA.
Measure: Number; unit: Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Participants | 21 | 23
Statistical Analysis 1: Comparison: Cohort I (DTG 50 mg OD); Test type: Superiority or Other; percentage of participants = 78, 95% CI 2-sided [58 to 91] — The estimated value represents the percentage of participants with HIV-1 RNA <400 c/mL or at least 0.7 log10 c/mL below their Baseline value at Day 11
Statistical Analysis 2: Comparison: Cohort II (DTG 50 mg BID); Test type: Superiority or Other; percentage of participants = 96, 95% CI [79 to 100] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Change From Baseline in Plasma HIV-1 RNA at Day 6 to 8, Day 11, Weeks 4, 12, 24, 48, 72, 96, From Week 108 Every 12 Weeks up to Study Completion
Description: Mean change from Baseline in Plasma HIV-1 RNA was assessed on Day 6 to 8, Day 11, and Weeks 4, 12, 24, 48, 72, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, and 264 using data of the observed cases. Study Day 1 was considered as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Day 6 to 8; Day 11; Weeks 4, 12, 24, 48, 72, 96, from 108 every 12 weeks up to study completion
Population: ITT-E Population. Only those participants available at the indicated time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Log10 copies/mL
  Day 6 to 8, n=27, 24 | -1.31 (0.71) | -1.40 (0.43)
  Day 11, n=27, 24 | -1.45 (0.77) | -1.76 (0.53)
  Week 4, n=26, 24 | -1.82 (1.03) | -2.06 (0.78)
  Week 12, n=22, 24 | -1.94 (1.14) | -2.30 (0.93)
  Week 24, n=18, 22 | -1.99 (1.08) | -2.50 (0.81)
  Week 48, n=15, 20 | -2.02 (1.07) | -2.63 (0.78)
  Week 72, n=14, 18 | -2.10 (1.03) | -2.71 (0.82)
  Week 96, n=13, 15 | -2.06 (1.13) | -2.58 (0.77)
  Week 108, n= 13, 17 | -1.95 (1.20) | -2.69 (0.82)
  Week 120, n= 11, 17 | -2.09 (1.15) | -2.67 (0.85)
  Week 132, n= 11, 17 | -1.83 (1.01) | -2.66 (0.86)
  Week 144, n= 12, 15 | -2.08 (1.29) | -2.62 (0.94)
  Week 156, n= 12, 15 | -2.04 (1.36) | -2.65 (0.77)
  Week 168, n= 11, 14 | -1.77 (1.26) | -2.72 (0.89)
  Week 180, n= 11, 10 | -1.76 (1.11) | -2.56 (0.82)
  Week 192, n= 9, 7 | -1.87 (1.16) | -2.51 (0.98)
  Week 204, n= 10, 6 | -1.76 (1.21) | -2.35 (0.71)
  Week 216, n= 9, 6 | -1.61 (1.08) | -2.35 (0.71)
  Week 228, n= 6, 4 | -1.79 (1.08) | -2.33 (0.90)
  Week 240, n= 7, 0 | -1.63 (1.13) | NA (NA) — Since 0 participants were analyzed, no data to present.
  Week 252, n= 4, 0 | -1.72 (1.07) | NA (NA) — Since 0 participants were analyzed, no data to present.
  Week 264, n= 1, 0 | -2.90 (NA) — As only 1 participant was analyzed; therefore, no SD to present. | NA (NA) — Since 0 participants were analyzed, no data to present.

3. Secondary Outcome: Number of Participants Who Achieved Plasma HIV-1 RNA <400 c/mL and <50 c/mL at Baseline and Weeks 4, 12, 24, 48, 72, and 96: TLOVR Analysis.
Description: The number of participants with plasma HIV-1 RNA <400 c/mL or <50 c/mL was assessed at Weeks 4, 12, 24, 48, 72, and 96 per the Food and Drug Administration's Time to Loss of Virological Response (TLOVR) algorithm. Using the TLOVR algorithm, participants are considered to have failed on therapy if they never achieved confirmed RNA levels below the threshold, if they had confirmed rebound of RNA above the threshold, if they made a non-permitted change in background regimen, or if they permanently discontinued investigational product for any reason.
Time Frame: Baseline; Weeks 4, 12, 24, 48, 72, and 96
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Participants
  Baseline, <50 c/mL | 0 | 0
  Week 4, <50 c/mL | 9 | 12
  Week 12, <50 c/mL | 13 | 16
  Week 24, <50 c/mL | 11 | 19
  Week 48, <50 c/mL | 9 | 17
  Week 72, <50 c/mL | 8 | NA — As of the data cut-off, Week 48 is the last time point which all participants in Cohort II would have had opportunity to reach if they had not discontinued prematurely. Only data to Week 48 were therefore analyzed using TLOVR.
  Week 96, <50 c/mL | 7 | NA — As of the data cut-off, Week 48 is the last time point which all participants in Cohort II would have had opportunity to reach if they had not discontinued prematurely. Only data to Week 48 were therefore analyzed using TLOVR.
  Baseline, <400 c/mL | 0 | 0
  Week 4, <400 c/mL | 16 | 17
  Week 12, <400 c/mL | 16 | 20
  Week 24, <400 c/mL | 14 | 20
  Week 48, <400 c/mL | 13 | 18
  Week 72, <400 c/mL | 12 | NA — As of the data cut-off, Week 48 is the last time point which all participants in Cohort II would have had opportunity to reach if they had not discontinued prematurely. Only data to Week 48 were therefore analysed using TLOVR.
  Week 96, <400 c/mL | 10 | NA — As of the data cut-off, Week 48 is the last time point which all participants in Cohort II would have had opportunity to reach if they had not discontinued prematurely. Only data to Week 48 were therefore analysed using TLOVR.

4. Secondary Outcome: Proportion of Participants Who Achieved Plasma HIV-1 RNA <400 c/mL and <50 c/mL From Week 48 Every 12 Weeks up to Study Completion
Description: The number of participants with plasma HIV-1 RNA <400 c/mL or <50 c/mL was assessed at Weeks 48, 72, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, and 264 using data of observed cases. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: From Week 48 every 12 weeks up to study completion
Population: ITT-E Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Percentage of Participants
  Week 48, <50 c/mL, n=15, 20 | 60 | 80
  Week 60, <50 c/mL, n=13, 18 | 69 | 94
  Week 72, <50 c/mL, n=14, 18 | 64 | 78
  Week 84, <50 c/mL, n=14, 18 | 57 | 78
  Week 96, <50 c/mL, n=13, 15 | 54 | 87
  Week 108, <50 c/mL, n=13, 17 | 54 | 88
  Week 120, <50 c/mL, n=11, 17 | 55 | 88
  Week 132, <50 c/mL, n=11, 17 | 55 | 82
  Week 144, <50 c/mL, n=12, 15 | 58 | 87
  Week 156, <50 c/mL, n=12, 15 | 67 | 93
  Week 168, <50 c/mL, n=11, 14 | 64 | 86
  Week 180, <50 c/mL, n=11, 10 | 64 | 100
  Week 192, <50 c/mL, n= 9, 7 | 67 | 100
  Week 204, <50 c/mL, n= 10, 6 | 50 | 100
  Week 216, <50 c/mL, n= 9, 6 | 56 | 100
  Week 228, <50 c/mL, n=6, 4 | 67 | 100
  Week 240, <50 c/mL, n=7,0 | 57 | NA — Since 0 participants were analyzed, no value to present.
  Week 252, <50 c/mL, n=4, 0 | 50 | NA — Since 0 participants were analyzed, no value to present.
  Week 264, <50 c/mL, n=1, 0 | 100 | NA — Since 0 participants were analyzed, no value to present.
  Week 48, <400 c/mL, n=15, 20 | 73 | 95
  Week 60,<400 c/mL, n=13, 18 | 92 | 100
  Week 72,<400 c/mL, n=14, 18 | 79 | 100
  Week 84,<400 c/mL, n=14, 18 | 71 | 94
  Week 96,<400 c/mL, n=13, 15 | 85 | 100
  Week 108,<400 c/mL, n=13,17 | 85 | 100
  Week 120,<400 c/mL, n=11, 17 | 82 | 94
  Week 132,<400 c/mL, n=11,17 | 82 | 94
  Week 144,<400 c/mL, n=12, 15 | 83 | 93
  Week 156,<400 c/mL, n=12, 15 | 75 | 100
  Week 168,<400 c/mL, n=11, 14 | 82 | 100
  Week 180,<400 c/mL, n=11, 10 | 73 | 100
  Week 192,<400 c/mL, n=9, 7 | 78 | 100
  Week 204,<400 c/mL, n=10, 6 | 70 | 100
  Week 216,<400 c/mL, n=9, 6 | 56 | 100
  Week 228,<400 c/mL, n=6, 4 | 67 | 100
  Week 240,<400 c/mL, n=7, 0 | 71 | NA — Since 0 participants were analyzed, no value to present.
  Week 252,<400 c/mL, n=4, 0 | 50 | NA — Since 0 participants were analyzed, no value to present.
  Week 264,<400 c/mL, n=1, 0 | 100 | NA — Since 0 participants were analyzed, no value to present.

5. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Day 11 and Weeks 4, 12, 24, 48, 72, 96, Week 108 Every 12 Weeks up to Study Completion
Description: Change from Baseline in CD4+ cell count was assessed at Day 11 and at Weeks 4, 12, 24, 48, 72, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, and 264 . Study Day 1 was considered as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Day 11; Weeks 4, 12, 24, 48, 72, 96, from Week 108 every 12 weeks up to study completion
Population: ITT-E Population. Only those participants available at the indicated time points were analyzed (represented by n=X in the category titles).
Measure: Median (Full Range); unit: cells per cubic millimeter (mm^3)
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
cells per cubic millimeter (mm^3)
  Baseline, n=27, 24 | 114 [44 to 227] | 202 [19 to 384]
  Day 11, n=27, 24 | 34 [2 to 71] | 14 [0 to 69]
  Week 4, n=27, 24 | 57 [33 to 108] | 35 [8 to 69]
  Week 12, n= 22, 24 | 84 [26 to 124] | 57 [8 to 103]
  Week 24, n=17, 22 | 78 [54 to 175] | 79 [17 to 147]
  Week 48, n=15, 20 | 102 [29 to 160] | 106 [45 to 245]
  Week 72, n=14, 18 | 163 [58 to 204] | 191.5 [80 to 277]
  Week 96, n=13, 15 | 142 [75 to 202] | 189 [75 to 280]
  Week 108, n=13, 17 | 124 [68 to 249] | 155 [91 to 276]
  Week 120, n=11, 17 | 221 [62 to 306] | 221 [135 to 314]
  Week 132, n=11, 17 | 97 [26 to 303] | 158 [129 to 384]
  Week 144, n=12, 15 | 121 [28 to 284] | 278 [113 to 340]
  Week 156, n=12, 15 | 212 [64 to 378] | 223 [131 to 309]
  Week 168, n=11, 13 | 97 [-102 to 365] | 271 [93 to 357]
  Week 180, n=11, 10 | 125 [55 to 327] | 224 [163 to 288]
  Week 192, n=10, 7 | 94 [61 to 291] | 343 [304 to 429]
  Week 204, n=10, 6 | 92 [47 to 364] | 264 [186 to 370]
  Week 216, n=9, 6 | 172 [48 to 416] | 252 [147 to 421]
  Week 228, n=7, 3 | 148 [66 to 357] | 417 [-12 to 633]
  Week 240, n=7, 0 | 158 [119 to 470] | NA [NA to NA] — Since 0 participants were analyzed, no data to present.
  Week 252, n=4, 0 | 157 [109 to 282] | NA [NA to NA] — Since 0 participants were analyzed, no data to present.
  Week 264, n=1, 0 | 560 [560 to 560] | NA [NA to NA] — Since 0 participants were analyzed, no data to present.

6. Secondary Outcome: Cmax, Cmin, and Ctau of DTG
Description: The maximum plasma concentration (Cmax), minimum plasma concentration (Cmin), and concentration at the end of a dosing interval (Ctau) of DTG were assessed at Day 10. Blood samples for pharmacokinetic (PK) assessments were collected at pre-dose (within 15 minutes prior to dose) and 2, 3, 4, 8, and 24 hours post-dose on Day 10 for DTG 50 mg OD and pre-dose (within 15 minutes prior to dose) and 2, 3, 4 and 8 hours post morning dose and 12 hours post evening dose for DTG 50 mg BID.
Time Frame: Day 10
Population: Pharmacokinetic (PK) Parameter Population: all participants who provided at least one evaluable PK concentration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (µg/mL)
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 25 | 23
Micrograms per milliliter (µg/mL)
  Cmax | 3.04 (38) | 5.41 (40)
  Ctau | 0.69 (91) | 2.72 (70)
  Cmin | 0.48 (136) | 2.61 (67)

7. Secondary Outcome: C0 Assessment of DTG
Description: The plasma DTG concentration immediately prior to dosing at steady state (C0) was assessed at Day 10, and Weeks 4 and 24. Blood samples for pharmacokinetic assessments were collected at pre-dose (within 15 minutes prior to dose).
Time Frame: Day 10; Weeks 4 and 24
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 25 | 23
µg/mL
  C0, Day 10 | 0.51 (139) | 3.20 (69)
  C0, Week 4 | 0.57 (100) | 2.55 (63)
  C0, Week 24 | 0.38 (114) | 2.38 (69)

8. Secondary Outcome: Tmax of DTG
Description: The tmax is defined as the time of occurrence of the maximum plasma concentration (Cmax). The tmax was assessed at Day 10. Blood samples for pharmacokinetic assessments were collected at pre-dose (within 15 minutes prior to dose) and 2, 3, 4, 8, and 24 hours post-dose on Day 10 for DTG 50 mg OD and pre-dose (within 15 minutes prior to dose) and 2, 3, 4 and 8 hours post morning dose and 12 hours post evening dose for DTG 50 mg BID.
Time Frame: Day 10
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 25 | 23
Hours | 2.97 [1.97 to 7.92] | 2.00 [0.00 to 7.87]

9. Secondary Outcome: AUC0-24 Assessment of DTG
Description: AUC is defined as the area under the DTG concentration-time curve as a measure of drug exposure. AUC(0-24) is defined as the area under the concentration-time curve from time zero (pre-dose) to 24 hours. AUC0-24 of DTG was assessed at Day 10. Blood samples for pharmacokinetic assessments were collected at pre-dose (within 15 minutes prior to dose) and 2, 3, 4, 8, and 24 hours post-dose on Day 10 for DTG 50 mg OD and pre-dose (within 15 minutes prior to dose) and 2, 3, 4 and 8 hours post morning dose and 12 hours post evening dose for DTG 50 mg BID.
Time Frame: Day 10
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms*hour per milliliter (µg*hr/mL
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 25 | 23
Micrograms*hour per milliliter (µg*hr/mL | 36.46 (53) | 93.36 (50)

10. Secondary Outcome: Number of Participants With the Indicated HIV-1 Associated Conditions, Excluding Recurrences
Description: The number of participants with post-Baseline emergent HIV-1 disease progression (Acquired immunodeficiency syndrome (AIDS) or death) was assessed per the Centers for Disease Control and Prevention (CDC) 1993 revised classification system for HIV infection and expanded surveillance case definition for AIDS among adolescents and adults. The CDC classifies HIV infection as Category A (participants with asymptomatic HIV infection, acute HIV infection with accompanying illness, or persistent generalized lymphadenopathy), Category B (participants with symptomatic non-AIDS condition, i.e., conditions that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or conditions are considered by physicians to have a clinical course or to require management that is complicated by HIV infection), and Category C (includes AIDS indicator conditions as defined by diagnostic or presumptive measures).
Time Frame: From the day of the first dose of study drug until study completion (median 605 days for Cohort I, median 1181 days for Cohort II)
Population: ITT-E Population. Participant may have more than one HIV associated condition. Each condition is counted only once per participant, regardless of recurrence.
Measure: Number; unit: Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Participants
  Category B, Candidiasis, oropharyngeal | 3 | 2
  Category B, Hairy leukoplakia, oral | 2 | 0
  Category B, Herpes Zoster | 2 | 0
  Category C, Herpes simplex | 1 | 0
  Category C, Candidiasis, esophageal | 0 | 1
  Category C, Cytomegalovirus retinitis | 0 | 1
  Category C, Kaposi's sarcoma | 1 | 0
  Category C, Lymphoma, Burkitt's | 0 | 1
  Category C, Lymphoma, immunoblastic | 1 | 0
  Death, Brain mass | 1 | 0
  Death, Completed suicide | 0 | 1
  Death, Febrile bone marrow aplasia | 1 | 0
  Death, Immunoblastic lymphoma | 1 | 0
  Death, Acute pulmonary oedema | 1 | 0
  Death, Anaemia | 0 | 1
  Death, Haemochromatosis | 0 | 1
  Death, Hepatic fibrosis | 0 | 1
  Other: Cryptosporidiosis, acute intestinal | 0 | 1
  Other: leukoplasia of both side of the tongue | 1 | 0

11. Secondary Outcome: Number of Participants With HIV-1 Associated Disease Progression With the Indicated Shifts to CDC Class C or Death
Description: The number of participants with HIV-1 disease progression (AIDS or death) was assessed per the CDC 1993 revised classification system for HIV infection and expanded surveillance case definition for AIDS among adolescents and adults. The CDC classifies HIV infection as Category A (participants with asymptomatic HIV infection, acute HIV infection with accompanying illness, or persistent generalized lymphadenopathy), Category B (participants with symptomatic non-AIDS condition, i.e., conditions that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or conditions are considered by physicians to have a clinical course or to require management that is complicated by HIV infection), and Category C (includes AIDS indicator conditions as defined by diagnostic or presumptive measures).
Time Frame: as for outcome 10
Population: ITT-E Population.
Measure: Number; unit: Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Participants
  From CDC class A to CDC class C | 0 | 2
  From CDC class B to CDC class C | 0 | 2
  From CDC class C to new CDC class C | 1 | 0
  From CDC Class A, B, or C to death | 3 | 2

12. Secondary Outcome: Number of Participants (Cumulative) With Protocol-defined Virological Failure (PDVF) at Day 11 and Weeks 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 84, 96, Week 108 Every 12 Weeks up to Study Completion
Description: PDVF is defined in relation to Baseline plasma HIV-1 RNA levels: at Day 11, a decrease of <0.7 log10 c/mL unless <400 c/mL; at Weeks 8 to <16, a decrease of <1.0 log10 c/mL unless <400 c/mL or an increase of >= 1.0 log10 c/mL from nadir; and at or after Week 16, ≥400 c/mL. PDVF at Day 11 was based on a single plasma HIV-1 RNA evaluation and did not require confirmation. Confirmation testing was required for visits at or after Week 8. For the combination treatment phase, all HIV-1 RNA samples that meet a criterion for suspected PDVF must be confirmed by a second measurement performed at least 1 week but not more than 4 weeks apart from the date of the original sample.
Time Frame: Day 11; Weeks 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 84, 96, from Week 108 every 12 weeks up to study completion
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Participants
  Day 11 | 6 | 1
  Week 8 | 7 | 3
  Week 12 | 9 | 3
  Week 16 | 10 | 5
  Week 20 | 10 | 5
  Week 24 | 12 | 5
  Week 32 | 12 | 5
  Week 40 | 12 | 5
  Week 48 | 13 | 5
  Week 60 | 13 | 5
  Week 72 | 14 | 6
  Week 84 | 15 | 6
  Week 96 | 16 | 6
  Week 108 | 16 | 6
  Week 120 | 16 | 6
  Week 132 | 16 | 6
  Week 144 | 16 | 7
  Week 156 | 16 | 7
  Week 168 | 16 | 7
  Week 180 | 16 | 7
  Week 192 | 16 | 7
  Week 204 | 16 | 7
  Week 216 | 17 | 7
  Week 228 | 18 | 7
  Week 240 | 18 | NA — No data were available for analysis from Cohort II at the time points.
  Week 252 | 18 | NA — No data were available for analysis from Cohort II at the time points.
  Week 264 | 18 | NA — No data were available for analysis from Cohort II at the time points.

13. Secondary Outcome: Number of Participants With the Indicated Genotypic Resistance at Baseline
Description: At Baseline, the integrase genotypic results were used to document resistance to raltegravir (RAL) and for the allocation of participants to one of two genotypic groups according to their RAL signature mutations to ensure a broad range of sensitivity to DTG. These results were not used to pre-define subgroup for analysis.
Time Frame: Baseline
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Participants
  Q148 + 2 | 3 | 2
  Q 148 + 1 | 4 | 8
  Mixture | 2 | 1
  Y143 | 12 | 6
  N155 | 4 | 6
  Other | 2 | 1

14. Secondary Outcome: Median Fold Change in Sensitivity to DTG by the Baseline (Day 1) IN Mutational Group
Description: Summary of median fold change in sensitivity to DTG by Integrase (IN) mutational group was assessed. The IN mutational group comprises of the following mutations: Q148 +2, Q148 +1, mixture (participants with virus containing more than one Y143, Q148 or N155 mutation at Day 1), Y143, N155, other (participants with virus having no mutations at codons 143, 148, or 155 at Day 1). Fold change (FC) is the fold change in 50% Inhibitory Concentration (IC50) relative to the wild-type control virus.
Time Frame: Baseline (Day 1)
Population: ITT-E Population
Measure: Median (Full Range); unit: Percentage
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Percentage
  Q148 + 2, n=3, 2 | 21 [14 to 35] | 4 [2.1 to 6.0]
  Q148 + 1, n=4, 8 | 5.5 [3.3 to 25] | 5.5 [4.1 to 8.2]
  Mixture, n=2, 1 | 7.8 [6.5 to 9.1] | 9.48 [9.48 to 9.48]
  Y143, n=12, 6 | 1.1 [0.6 to 1.4] | 1.2 [0.92 to 1.8]
  N155, n=4, 6 | 1.8 [1.5 to 5.1] | 2.3 [1.3 to 4.0]
  Other, n=2, 1 | 1.2 [0.9 to 1.5] | 0.87 [0.87 to 0.87]

15. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent Integrase (IN) Mutations Detected at the Time of Protocol-defined Virologic Failure (PDVF) as a Measure of Genotypic Resistance
Description: An analysis of changes at specific amino acids in the IN coding region associated with resistance to raltegravir, elvitegravir, or DTG was performed at Day 1 and at the time of PDVF. PDVF is defined in relation to Baseline plasma HIV-1 RNA levels: at Day 11, a decrease of <0.7 log10 c/mL unless <400 c/mL; at Weeks 8 to <16, a decrease of <1.0 log10 c/mL unless <400 c/mL or an increase of >= 1.0 log10 c/mL from nadir; and at or after Week 16, ≥400 c/mL. PDVF at Day 11 was based on a single plasma HIV-1 RNA evaluation and did not require confirmation. Confirmation testing was required for visits at or after Week 8. For the combination treatment phase, all HIV-1 RNA samples that meet a criterion for suspected PDVF must be confirmed by a second measurement performed at least 1 week but not more than 4 weeks apart from the date of the original sample.
Time Frame: From Baseline (Day 1) until study completion (median 605 days for Cohort I, median 1181 days for Cohort II)
Population: On-treatment Genotypic Resistance Population: all ITT-E participants who met the criteria for protocol-defined virological failure (PDVF)
Measure: Number; unit: Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 18 | 7
Participants
  Any | 11 | 5
  E138T | 0 | 1
  N155H | 3 | 4
  T97A | 2 | 0
  E92E/Q | 0 | 1
  G140S | 3 | 0
  L74I/M | 1 | 0
  Q148H | 2 | 0
  E138E/A | 1 | 0
  E138E/K | 1 | 2
  L74I/M/I | 1 | 0
  L74M | 1 | 0
  L74I | 1 | 0
  T97T/A | 0 | 2
  Q148R | 1 | 0
  S147G | 3 | 0
  E92E/V | 0 | 1
  L68L/I | 1 | 0

16. Secondary Outcome: Number of Participants With the Indicated Fold Increase in DTG FC (Fold Change in IC50 Relative to Wild-type Virus) Between Baseline and the Time of PDVF, as a Measure of Post-Baseline Phenotypic Resistance
Description: The FC in IC50 (50% inhibitory concentration) for DTG relative to wild-type virus was determined for virus isolated at Baseline and at the time of PDVF.The number of participants with the indicated change (ratio) in the two values at the time of PDVF is presented. PDVF is defined in relation to Baseline plasma HIV-1 RNA levels: at Day 11, a decrease of <0.7 log 10 c/mL unless <400 c/mL; at Weeks 8 to <16, a decrease of <1.0 log 10 c/mL unless <400 c/mL or an increase of >=1.0 log 10 c/mL from nadir; and at or after Week 16, ≥400 c/mL . PDVF at Day 11 was based on a single plasma HIV-1 RNA evaluation and did not require confirmation. Confirmation testing was required for visits at or after Week 8. For the combination treatment phase, all HIV-1 RNA samples that meet a criterion for suspected PDVF must be confirmed by a second measurement performed at least 1 week but not more than 4 weeks apart from the date of original sample.
Time Frame: From Baseline (Day 1) until study completion (median 605 days for Cohort I, median 1181 days for Cohort II)
Population: PDVF Phenotypic Resistance Populations: all participants in the ITT-E Population with available on-treatment phenotypic resistance data at the time of PDVF failure. Only participants with both Baseline and PDVF time-point DTG phenotypic data were considered for analysis.
Measure: Number; unit: Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 17 | 7
Participants
  <1 fold | 3 | 0
  1-<2 fold | 4 | 2
  2-<4 fold | 1 | 0
  4-<8 fold | 1 | 2
  >=8 fold | 8 | 3

17. Secondary Outcome: Number of Participants With the Indicated Grade 3 and Grade 4 Clinical Chemistry Toxicities
Description: Hematology and clinical chemistry data were summarized according to Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, dated December 2004. Grade 1, Mild; Grade 2, Moderate; Grade 3, Severe; Grade 4, Potentially life-threatening. Data are presented for only those parameters for which an increase to Grade 3 or Grade 4 occurred. The Grade 3 and Grade 4 clinical chemistry toxicities included: Albumin, Alkaline Phosphatase, Amylase, Aspartate Amino Transferase, Carbon dioxide content/Bicarbonate, Creatinine, Creatinine Clearance, Hypercalcemia, Hyperglycaemia, Hyperkalemia, Hypernatremia, Hypocalcemia, Hypoglycaemia, Hypokalemia, Hyponatremia, LDL Cholesterol, Magnesium, Phosphorus inorganic, and Total Bilirubin, Alanine Amino Transferase, Calcium, Chloride, Cholesterol, Creatine Kinase, Direct Bilirubin, Glucose, High Density Lipid (HDL), Cholesterol direct, Lipase, Potassium, Sodium, Total Cholesterol, Triglycerides, Urea/Blood Urine Nitrogen.
Time Frame: From start of study treatment until the end of treatment visit for each participant, up to Week 264 for Cohort I and up to Week 228 for Cohort II
Population: Safety Population: all participants that took at least one dose of DTG
Measure: Number; unit: Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Participants
  Albumin, Grade 3 | 0 | 0
  Albumin, Grade 4 | 0 | 0
  Alkaline Phosphatase, Grade 3 | 0 | 0
  Alkaline Phosphatase, Grade 4 | 0 | 0
  Amylase, Grade 3 | 1 | 2
  Amylase, Grade 4 | 1 | 0
  Aspartate Amino Transferase, Grade 3 | 0 | 0
  Aspartate Amino Transferase, Grade 4 | 0 | 0
  Carbon dioxide content/Bicarbonate, Grade 3 | 0 | 0
  Carbon dioxide content/Bicarbonate, Grade 4 | 0 | 0
  Creatinine, Grade 3 | 0 | 0
  Creatinine, Grade 4 | 0 | 0
  Creatinine Clearance, estimated, Grade 3 | 0 | 0
  Creatinine Clearance, estimated, Grade 4 | 0 | 0
  Hypercalcemia, Grade 3 | 0 | 0
  Hypercalcemia, Grade 4 | 0 | 0
  Hyperglycaemia, Grade 3 | 0 | 0
  Hyperglycaemia, Grade 4 | 0 | 0
  Hyperkalemia, Grade 3 | 0 | 0
  Hyperkalemia, Grade 4 | 0 | 0
  Hypernatremia, Grade 3 | 1 | 0
  Hypernatremia, Grade 4 | 0 | 0
  Hypocalcemia, Grade 3 | 0 | 0
  Hypocalcemia, Grade 4 | 0 | 0
  Hypoglycaemia, Grade 3 | 1 | 0
  Hypoglycaemia, Grade 4 | 0 | 1
  Hypokalemia, Grade 3 | 0 | 0
  Hypokalemia, Grade 4 | 0 | 0
  Hyponatremia, Grade 3 | 0 | 0
  Hyponatremia, Grade 4 | 0 | 0
  LDL Cholesterol, Grade 3 | 2 | 1
  LDL Cholesterol, Grade 4 | 0 | 0
  Magnesium, Grade 3 | 0 | 0
  Magnesium, Grade 4 | 0 | 0
  Phosphorus inorganic, Grade 3 | 4 | 3
  Phosphorus inorganic, Grade 4 | 0 | 0
  Total Bilirubin, Grade 3 | 0 | 2
  Total Bilirubin, Grade 4 | 0 | 1
  Alanine Amino Transferase ,Grade 3 | 0 | 1
  Alanine Amino Transferase ,Grade 4 | 0 | 0
  Calcium,Grade 3 | 0 | 0
  Calcium,Grade 4 | 0 | 0
  Chloride,Grade 3 | 0 | 0
  Chloride,Grade 4 | 0 | 0
  Cholesterol,Grade 3 | 1 | 1
  Cholesterol,Grade 4 | 0 | 0
  Creatine Kinase,Grade 3 | 0 | 0
  Creatine Kinase,Grade 4 | 0 | 0
  Direct Bilirubin,Grade 3 | 0 | 0
  Direct Bilirubin,Grade 4 | 0 | 0
  Glucose,Grade 3 | 1 | 0
  Glucose,Grade 4 | 0 | 1
  HDL Cholesterol direct,Grade 3 | 0 | 0
  HDL Cholesterol direct,Grade 4 | 0 | 0
  Lipase,Grade 3 | 2 | 3
  Lipase,Grade 4 | 1 | 1
  Potassium,Grade 3 | 0 | 0
  Potassium,Grade 4 | 0 | 0
  Sodium,Grade 3 | 1 | 0
  Sodium,Grade 4 | 0 | 0
  Total Cholesterol/HDLratio, Grade 3 | 0 | 0
  Total Cholesterol/HDLratio, Grade 4 | 0 | 0
  Triglycerides,Grade 3 | 0 | 2
  Triglycerides,Grade 4 | 0 | 0
  Urea/BUN,Grade 3 | 0 | 0
  Urea/BUN,Grade 4 | 0 | 0

18. Secondary Outcome: Number of Participants With the Indicated Grade 3 and Grade 4 Hematological Toxicities
Description: Hematology and clinical chemistry data were summarized according to Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, dated December 2004. Grade 1, Mild; Grade 2, Moderate; Grade 3, Severe; Grade 4, Potentially life-threatening. Data are presented for only those parameters for which an increase to Grade 3 or Grade 4 occurred. The Grade 3 and Grade 4 hematological toxicities included: Hemoglobin, Platelet Count, Total Neutrophils, and White Blood Cell count.
Time Frame: as for outcome 17
Population: Safety Population: all participants that took at least one dose of DTG
Measure: Number; unit: Participants
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Number analyzed (Participants) | 27 | 24
Participants
  Hemoglobin, Grade 3 | 0 | 1
  Hemoglobin, Grade 4 | 0 | 0
  Platelet count, Grade 3 | 0 | 0
  Platelet count, Grade 4 | 0 | 0
  Total Neutrophils, Grade 3 | 0 | 0
  Total Neutrophils, Grade 4 | 0 | 2
  White Blood Cell count, Grade 3 | 0 | 0
  White Blood Cell, Grade 4 | 0 | 1

ADVERSE EVENTS:
Time Frame: SAEs, non-serious AEs and laboratory toxicities were collected from start of study treatment until the end of treatment visit for each participant, up to Week 264 for Cohort I and up to Week 228 for Cohort II.
Description: SAEs and non-serious AEs were collected in the Safety Population, comprised of all participants that took at least one dose of DTG.
Arm/Group | Cohort I (DTG 50 mg OD) | Cohort II (DTG 50 mg BID)
Serious Adverse Events (participants affected / at risk) | 10/27 | 11/24
Other Adverse Events (participants affected / at risk) | 25/27 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I (DTG 50 mg OD) (N=27) | Cohort II (DTG 50 mg BID) (N=24)
Gastroenteritis viral (Infections and infestations) | 0 | 1
Neurosyphilis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Body fat disorder (Metabolism and nutrition disorders) | 1 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Immunoblastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain mass (Nervous system disorders) | 1 | 0
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Anogenital dysplasia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Cryoglobulinaemia (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 1 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I (DTG 50 mg OD) (N=27) | Cohort II (DTG 50 mg BID) (N=24)
Diarrhoea (Gastrointestinal disorders) | 8 | 9
Bronchitis (Infections and infestations) | 6 | 7
Pyrexia (General disorders) | 3 | 7
Asthenia (General disorders) | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Headache (Nervous system disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Fatigue (General disorders) | 0 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Rhinitis (Infections and infestations) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Backpain (Musculoskeletal and connective tissue disorders) | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Influenza like illness (General disorders) | 0 | 2
Injection site reaction (General disorders) | 0 | 2
Lipase increased (Investigations) | 0 | 3
Oedema peripherial (General disorders) | 4 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sinusitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 5
Urinary tract infection (Infections and infestations) | 0 | 3
Vertigo (Ear and labyrinth disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Herpes virus infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 3 | 0
Oral herpes (Infections and infestations) | 3 | 0
Tooth abscess (Infections and infestations) | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 2
Defaecation urgency (Gastrointestinal disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2
Gastroenteritis viral (Infections and infestations) | 3 | 0
Ear infection (Infections and infestations) | 2 | 0
Genital herpes (Infections and infestations) | 2 | 0
Otitis media (Infections and infestations) | 2 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 2 | 0
Malaise (General disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sciatica (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 0 | 2
Dysaesthesia (Nervous system disorders) | 2 | 0
Anxiety (Nervous system disorders) | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 2 | 0
Weight decreased (Investigations) | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 2
Seasonal allergy (Immune system disorders) | 2 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Hypertension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.